CLINICAL TRIAL: NCT06654960
Title: A Single Center, Open-label, Single Cohort, Fixed Sequence Trial, Investigating the Influence of HRS9531 Injection on Pharmacokinetics of Metformin in Healthy Subjects
Brief Title: Influence of HRS9531 on Pharmacokinetics of Metformin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS9531-106
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: HRS9531 injection; Drug: Metformin Hydrochloride tablets

INTERVENTIONS:
Drug: HRS9531 injection — HRS9531 injection single dose.
Drug: Metformin Hydrochloride tablets — Metformin Hydrochloride tablets 500mg.

SUMMARY:
The purpose of this study is to evaluate the influence of HRS9531 injection on pharmacokinetics of metformin in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the trial procedures and possible adverse events, be able and willing to provide a written informed consent;
2. Male subjects aged 18-45 years on the date of signing informed consent (inclusive);
3. Body weight ≥50 kg, body mass index (BMI) within the range of 20.0-30.0 kg/m2 (inclusive);
4. HbA1c<6.0%.

Exclusion Criteria:

1. Chronic or severe medical history of the respiratory system, circulatory system, digestive system, urinary system, blood system, endocrine system, immune system, nervous system, mental system, etc., or those with existing systemic diseases mentioned above, and judged by the investigator to be unsuitable to participate in this study;
2. Obvious gastric emptying abnormalities or gastrointestinal diseases in the past, or had undergone gastrointestinal surgery (except for gastrointestinal polyps, appendix, and haemorrhoidectomy)
3. Past history or family history of medullary thyroid cancer or multiple endocrine neoplasia type 2 (MEN2), a history of pancreatitis or symptomatic gallbladder stones;
4. Surgery within 6 months prior to dosing, planned to undergo surgery during the study period;
5. Participation in clinical trials of any drug or medical device in the 3 months or 5 half-lives, whichever longer, prior to dosing;
6. Blood donation history or blood loss ≥400 mL within 3 months or ≥200 mL within 1 month before dosing, or received blood transfusion within 3 months before dosing;
7. Allergic constitution includes severe drug allergy or history of drug allergy;
8. Hepatitis B surface antigen (HBsAg), HIV antibody, hepatitis C virus antibody (HCVAb), treponema pallidum specific antibody detection, positive;
9. Abnormal laboratory test results or abnormal examinations considered unsuitable to participate in this trial;
10. History of hypoglycaemia;
11. The investigator considers that the subject has any other factors that would make it inappropriate to participate in this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2024-12-26 (Actual)

PRIMARY OUTCOMES:
Area under the concentration versus time curve (AUC) of metformin from dosing time (0) to tau (dosing interval) (AUCtau) after 3.5 days. | Start of treatment up to 12 hours.

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) of metformin after 3.5 days of treatment. | Start of Treatment up to 30 hours.
Maximum concentration (Cmax) of metformin after 3.5 days of treatment. | Start of Treatment up to 30 hours.
Area under the concentration versus time curve of metformin from 0 to the time of the last measurable (positive) concentration (AUC0-t) after 3.5 days of treatment. | Start of Treatment up to 30 hours.
Area under the concentration versus time curve of metformin from 0 to infinity (AUC0-inf) after 3.5 days of treatment. | Start of Treatment up to 30 hours.
Terminal half-life (t1/2) of metformin after 3.5 days of treatment. | Start of Treatment up to 30 hours.
Clearance (CL/F) of metformin after 3.5 days of treatment. | Start of Treatment up to 30 hours.
Apparent volume of distribution (VzF) of metformin after 3.5 days of treatment. | Start of Treatment up to 30 hours.
Time to maximum concentration (Tmax) of HRS9531. | Start of Treatment up to 504 hours.
Maximum concentration (Cmax) of HRS9531. | Start of Treatment up to 504 hours.
Area under the concentration versus time curve of HRS9531 from 0 to the time of the last measurable (positive) concentration (AUC0-t). | Start of Treatment up to 30 hours.
Area under the concentration versus time curve of HRS9531 from 0 to infinity (AUC0-inf). | Start of Treatment up to 504 hours.
Terminal half-life (t1/2) of HRS9531. | Start of Treatment up to 504 hours.
Clearance (CL/F) of HRS9531. | Start of Treatment up to 504 hours.
Apparent volume of distribution (VzF) of HRS9531. | Start of Treatment up to 504 hours.
Incidence and severity of adverse events. | Screening period up to 42 days.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided